CLINICAL TRIAL: NCT00005937
Title: A Phase II Study of Antithymocyte Globulin (ATG) and Cyclosporine to Treat the Cytopenia of Myelodysplastic Syndrome (MDS)
Brief Title: Antithymocyte Globulin and Cyclosporine to Treat Myelodysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neal Young, M.D. (NIH)
Responsible Party: Sponsor-Investigator, Neal Young, M.D., NHLBI Hematolgy Branch Chief, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000169; 00-H-0169 (Other: NIH NHLBI)
Record Dates: First submitted 2000-07-06; First posted 2000-07-07 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; Immunosuppression; ATG; Cyclosporine; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antithymocyte globulin & cyclosporine (Experimental): Myelodysplastic syndromes (MDS) subjects will be treated with Anti-thymocyte Globulin (ATG) and cyclosporine (CsA). The subjects will receive ATG at a dose of 40mg/kg orally on days 1-4 in combination with oral prednisone at a dose of 1mg/kg/day on day one. The prednisone will be tapered on day 10. The taper schedule will be every two days over a total of eight days (days 10-17). Drug the ATG administration the subjects will receive at least 4 units of platelets daily for platelet counts less than 20,000/ microliters. Cyclosporine (CsA) will be started on day 14 at a dose of 5mg/kg twice daily with dose adjustments based on drug levels (target 200-400 ng/ml). Cyclosporine therapy will be continued for six months.
  Interventions: Drug: Antithymocyte globulin; Drug: Cyclosporine

INTERVENTIONS:
Drug: Antithymocyte globulin — Antithymocyte globulin (ATG) intravenous infusion: 40mg/kg/day. Infusion over 6 hours on day 1-4.
Drug: Cyclosporine — Cyclosporine (CsA) intravenous infusion: 5mg/kg. Infusion on day 14 administered twice a day.

SUMMARY:
This study will determine the safety and effectiveness of a combination of the immune-suppressing drugs antithymocyte globulin (ATG) and cyclosporine for treating myelodysplasia, a disorder of low blood cell counts. It will: evaluate whether this drug combination can increase blood counts in patients and reduce their need for transfusions; compare survival of patients who respond to ATG and cyclosporine treatment with those who do not respond; and determine the side effects of the treatment.

Myelodysplasia is thought to result from an immune system abnormality in which cells called lymphocytes attack the marrow's blood-forming cells. The resulting deficiencies of platelets and red and white blood cells cause anemia, susceptibility to infections, and easy bruising and bleeding. Various therapies, such as blood transfusions for anemia and bleeding, antibiotics for infection, chemotherapy and bone marrow transplantation are used to treat myelodysplasia, but all have disadvantages and some carry serious risks.

Patients 18 years of age and older with myelodysplasia may be eligible for this study. Candidates will be screened with a physical examination and medical history, blood tests, chest X-ray, electrocardiogram and bone marrow biopsy (removal of a marrow sample from the hipbone for microscopic examination).

DETAILED DESCRIPTION:
Participants will be admitted to the NIH Clinical Center for the first 10 to 14 days of treatment and will then continue therapy on an outpatient basis. They will undergo the following tests and procedures:

* Placement of central line-An intravenous (IV) catheter (flexible tube inserted into a vein) is placed in a large vein of the neck, chest or arm. Medicines are delivered through this line and blood samples are drawn from it.
* ATG skin testing- ATG is injected under the skin to check for sensitization to horse serum, from which the drug is derived.
* ATG treatment-Four doses of ATG are given through the IV line on each of 4 consecutive days. Prednisone is taken by mouth beginning the first day of ATG therapy and continuing for a total of 17 days. This drug is given to reduce the side effects of ATG, such as fever, skin rash and chills.
* Cyclosporine treatment- Cyclosporine capsules are taken by mouth twice a day for at least 6 months.

During hospitalization, blood will be drawn daily for blood counts and other tests. Upon the patient's discharge after 10 days, the referring physician will do blood tests weekly during the first month of treatment and then every 2 weeks for the rest of the time the patient is taking cyclosporine. Dosages of this drug may be adjusted depending on the test results. Patients will be evaluated at the NIH Clinical Center at 3-month intervals for the first year, then every 6 months for the next 3 years and then at yearly intervals. A blood sample will be drawn at each visit. Bone marrow biopsies will be done at 6-month intervals for the first 3 years after treatment.

A growing body of laboratory and clinical evidence suggests that the cytopenia of MDS is at least partly a result of cytotoxic T cell activity. Treatments to abrogate T cell activity such as anti-thymocyte globulin alone and cyclosporine alone have demonstrated varying degrees of success in alleviating the cytopenia of MDS. A response to such therapy in MDS is associated with improved survival. Experience with aplastic anemia suggests that the combination of these two agents should be more effective in suppressing cytotoxic T cell activity and alleviating cytopenia. This protocol proposes using the combination of antithymocyte globulin (ATG) and cyclosporine (CSA) to treat the cytopenia of MDS, in an effort to improve the response rate to immunosuppressive therapy in this disease.

ELIGIBILITY:
INCLUSION CRITERIA:

* MDS of refractory anemia (RA), refractory anemia with ring sideroblasts (RARS) & refractory anemia with excess blasts (RAEB) sub-types
* Off all other treatments (except G-CSF (granulocyte colony stimulating factor), and transfusion support and related medications) for at least four weeks.
* G-CSF can be used before, during and after the protocol treatment for patients with documented neutropenia (less than 500/uL) as long as they meet the criteria for anemia and/or thrombocytopenia as stated above.
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* High or intermediate predicted probability of response

EXCLUSION CRITERIA:

* MDS of FAB sub-group chronic myelomonocytic leukemia (CMML)
* Transformation to acute leukemia (FAB sub-group RAEB-T, ie., greater than 20% blasts in marrow aspirate)
* Hypoplastic marrow without one major or two minor criteria
* Treatment with growth factors (except for G-CSF) or cyclosporine within 4 weeks prior to entry to protocol
* ECOG performance status of greater than 2
* Active uncontrolled infection
* Current pregnancy, or unwilling to take oral contraceptives if of childbearing potential
* Patients for whom bone marrow transplant is indicated as standard therapy (age less than fifty-five with a fully-matched sibling donor)
* Age less than18 years
* Not able to give informed consent
* HIV positive patients
* Active malignant disease (excluding basal cell carcinoma)
* Serum creatinine greater than 2mg/dl
* Patients who are moribund or patients with concurrent hepatic, renal, cardiac, metabolic, or any disease of such severity that death within 3 months is likely
* Low predicted probability of response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2000-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Young, MD, Principal Investigator — NIH National Heart, Lung, and Blood Institute
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bynoe AG, Scott CS, Ford P, Roberts BE. Decreased T helper cells in the myelodysplastic syndromes. Br J Haematol. 1983 May;54(1):97-102. doi: 10.1111/j.1365-2141.1983.tb02071.x. PMID 6221751
- [Background] Porta F, Facchetti F, Tettoni K, Laffranchi MG, Arrighini A, Ugazio AG. Myelodysplastic syndrome in an infant: induction of remission by cyclosporin. Lancet. 1998 Nov 14;352(9140):1600-1. doi: 10.1016/s0140-6736(05)61048-3. No abstract available. PMID 9843114
- [Background] Nydegger UE. Suppressive and substitutive immunotherapy: an essay with a review of recent literature. Immunol Lett. 1985;9(4):185-90. doi: 10.1016/0165-2478(85)90031-8. No abstract available. PMID 3888832
- [Derived] Mehta SD, Moses S, Agot K, Maclean I, Odoyo-June E, Li H, Bailey RC. Medical male circumcision and herpes simplex virus 2 acquisition: posttrial surveillance in Kisumu, Kenya. J Infect Dis. 2013 Dec 1;208(11):1869-76. doi: 10.1093/infdis/jit371. Epub 2013 Jul 30. PMID 23901089
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2000-H-0169.html

RESULTS

PARTICIPANT FLOW:
Groups:
- MDS Subjects Treated With ATG & CsA: Myelodysplastic syndromes (MDS) subjects will be treated with Anti-thymocyte Globulin (ATG) and cyclosporine (CsA). The subjects will receive ATG at a dose of 40mg/kg orally on days 1-4 in combination with oral prednisone at a dose of 1mg/kg/day on day one. The prednisone will be tapered on day 10. The taper schedule will be every two days over a total of eight days (days 10-17). Drug the ATG administration the subjects will receive at least 4 units of platelets daily for platelet counts less than 20,000/ microliters. Cyclosporine (CsA) will be started on day 14 at a dose of 5mg/kg twice daily with dose adjustments based on drug levels (target 200-400 ng/ml). Cyclosporine therapy will be continued for six months.
Period: Overall Study
Arm/Group | MDS Subjects Treated With ATG & CsA
Started | 42
Completed | 37
Not Completed | 5
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Groups:
- MDS Subjects Treated With ATG and CsA: Myelodysplastic syndromes (MDS) subjects will be treated with Antithymocyte Globulin (ATG) and cyclosporine (CsA). The subjects will receive ATG at a dose of 40mg/kg orally on days 1-4 in combination with oral prednisone at a dose of 1mg/kg/day on day one. The prednisone will be tapered on day 10. The taper schedule will be every two days over a total of eight days (days 10-17). Drug the ATG administration, the subjects will receive at least 4 units of platelets daily for platelet counts less than 20,000/ microliters. Cyclosporine (CsA) will be started on day 14 at a dose of 5mg/kg twice daily with dose adjustments based on drug levels (target 200-400 ng/ml). Cyclosporine therapy will be continued for six months.
Arm/Group | MDS Subjects Treated With ATG and CsA
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell Transfusion Independence
Description: Red blood cell transfusion independence was documented as time from last transfusion of red cells to last day of transfusion free follow-up. Independence or response to the intervention was assessed by weekly blood counts. Transfusion independence was defined as no transfusion requirement for a 3 month period. Complete hematologic response is defined as the normalization of affected cells lines and less than 5% marrow blasts present. Partial hematologic response is defined as greater than 50% improvement from baseline to normal levels of all cell counts and greater than 50% decrease in marrow blasts.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- MDS Subjects Treated With ATG and CsA: Myelodysplastic syndromes (MDS) subjects will be treated with Anti-thymocyte Globulin (ATG) and cyclosporine (CsA). The subjects will receive ATG at a dose of 40mg/kg orally on days 1-4 in combination with oral prednisone at a dose of 1mg/kg/day on day one. The prednisone will be tapered on day 10. The taper schedule will be every two days over a total of eight days (days 10-17). Drug the ATG administration the subjects will receive at least 4 units of platelets daily for platelet counts less than 20,000/ microliters. Cyclosporine (CsA) will be started on day 14 at a dose of 5mg/kg twice daily with dose adjustments based on drug levels (target 200-400 ng/ml). Cyclosporine therapy will be continued for six months.
Arm/Group | MDS Subjects Treated With ATG and CsA
Number analyzed (Participants) | 37
participants
  Complete hematologic response | 6
  Partial hematologic response | 10
  No hematologic response | 21

ADVERSE EVENTS:
Arm/Group | MDS Subjects Treated With ATG and CsA
Serious Adverse Events (participants affected / at risk) | 11/42
Other Adverse Events (participants affected / at risk) | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDS Subjects Treated With ATG and CsA (N=42)
Death (Infections and infestations) | 7 (7)
Hospitalization pulmonary related (General disorders) | 2 (2)
Hospitalization cardiac related (Cardiac disorders) | 1 (1)
Hospitalization (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.76% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDS Subjects Treated With ATG and CsA (N=42)
Toxicity with disease progression (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes